CLINICAL TRIAL: NCT01572376
Title: Treatment of Pressure Ulcers With Autologous Bone Marrow Stem Cells in Spinal Cord Injury Patients.Phase I/II Study.
Brief Title: Autologous Bone Marrow Stem Cells in Pressure Ulcer Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Central de Asturias (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HUCentralAsturias
Record Dates: First submitted 2012-03-28; First posted 2012-04-06 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Type IV Pressure Ulcers; Chronic Wounds; Spinal Cord Injury
Keywords: Pressure ulcers; Chronic wounds; Spinal cord injury patients; Bone marrow; Mononuclear; Debridement
MeSH Terms: conditions — Spinal Cord Injuries; Pressure Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bone marrow stem cells (Experimental): Bone marrow was obtained by posterosuperior iliac crest aspiration under topical anesthesia. Mononuclear cells were isolated by Ficoll density gradient and will be resuspended in heparinized isotonic saline for infusion into the wound.
  Interventions: Procedure: Infusion of autologous bone marrow stem cells after wound debridement.

INTERVENTIONS:
Procedure: Infusion of autologous bone marrow stem cells after wound debridement. — Cleaning of the wound with heparinized saline, cell infusion and closing with suture.

SUMMARY:
The aim of the study is to determine the safety and feasibility of an autologous mononuclear stem cells infusion in pressure ulcers of paraplegic patients; and moreover, to evaluate the efficacy of the treatment.

DETAILED DESCRIPTION:
Taking into account the encouraging results obtained in the treatment of non-healing chronic wounds using bone marrow cells Given that treatment strategies for pressure ulcers can be both costly and complex, in this study we examine the possibility of improving pressure ulcer healing using stem cell therapy.

ELIGIBILITY:
Inclusion Criteria:

* Type IV ulcer pressures of more than 4 months topical treatment without response
* No option for conventional surgery
* Age range of 18-75 years old

Exclusion Criteria:

* Patients out of inclusion age range
* Patients with evidences of mental illness
* Patients with evidences of previous alcohol or drugs dependencies
* Pregnant women
* Patients with present or previous malignant disease during the last 5 years, except for basal cell carcinoma

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Absence of adverse effects during timeframe as infections or complications related with the intervention. | Six months
  The proposed trial will involve the recruitment of a total of 30 patients. The cells will be collected via bone marrow sampling. The aspirate will centrifuged on a Ficoll density gradient to isolate mononuclear cells, wich will be resuspended in heparinized isotonic saline for infusion into the area of the wound. Assessment of adverse events will be by wound examination and laboratory (microbiological)parameters

SECONDARY OUTCOMES:
Improvement and closure of the pressure ulcer | One year
  The closure of the ulcer will be assessed by NMR and physical examination

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias, Spain

REFERENCES:
- [Background] Sarasua JG, Lopez SP, Viejo MA, Basterrechea MP, Rodriguez AF, Gutierrez AF, Gala JG, Menendez YM, Augusto DE, Arias AP, Hernandez JO. Treatment of pressure ulcers with autologous bone marrow nuclear cells in patients with spinal cord injury. J Spinal Cord Med. 2011;34(3):301-7. doi: 10.1179/2045772311Y.0000000010. PMID 21756569